CLINICAL TRIAL: NCT06325436
Title: Accuracy of Simple Objective Scores in Prediction of Short-Term Outcome Among Cirrhotic Patients With Variceal Bleeding
Brief Title: Objective Scores in Variceal Bleeding
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rawnaa Hosny Ammar, Resident doctor, Assiut University
Other Study IDs: scores in variceal bleeding
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Variceal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the prognostic performance of the ALBI associated scores (ALBI, PALBI and INR-ALBI score) and new MELD .3 in predicting the short-term outcomes (early re-bleeding and early mortality) of patients with cirrhosis presenting with acute variceal bleeding, comparable to the CTP and MELD and MELD Na scores.

DETAILED DESCRIPTION:
Acute variceal bleeding is the most common feature of decompensation in patients with cirrhosis and one of the life-threatening complications, causing significant morbidity and mortality in patients with cirrhosis 2,3.

Although much progress has been made in diagnosis and treatment the 6-week mortality rate remains high, ranging from 10 to 20%, mainly due to failure to control bleeding in the first days 4-5.

It is therefore critical to develop a prognostic method for patients with acute variceal bleeding to determine the risk of re-bleeding 6 and resistance to standard treatment (accounting for 20-30%) 7 and death to adopt more aggressive treatment measures.

Many existing scoring systems have been used to evaluate the prognosis of patients with variceal bleeding, but none of them are targeted: including the Child-Pugh score, Model for End-Stage Liver Disease (MELD), and MELD-Na, clinical Rockall score (CRS), AIMS65 score (AIMS65), and Glasgow-Blatchford score (GBS) 9-11 However, these scores have the limitation that some information is subjective, and they use several tests that are less specific for liver disease, meaning that the best method to stratify risk of re-bleeding and morality among cirrhotic patients is still not clear.

In recent years, some new scores have been introduced. One of these scoring systems is the serum albumin and total bilirubin (ALBI) score that was developed to assess outcome in patients with hepatocellular carcinoma (HCC) and primary biliary cholangitis.

ALBI grade is a simple score derived from an easily accessible without using those factors evaluated subjectively (such as ascites and encephalopathy)14 and some studies suggest that it may provide better/similar prognostic performance compared with other well established prognostic scores like CTP score, MELD score 15.

The platelet-albumin-bilirubin (PALBI) score16 was initially used for the assessment of patients with HCC undergoing resection or ablation and later has been used as a predictor of mortality in patients with cirrhosis related complications 17.

PALBI score on admission is a good prognostic indicator for patients with acute variceal bleeding and predicts early mortality and rebleeding. The PALBI score performed better in predicting short-term outcome and the incidence of rebleeding compared with the other 4 scoring systems for acute variceal bleeding 18 .

Another simple score, the international normalized ratio-albumin-bilirubin (INR-ALBL) score, to predict rebleeding in patients with esopho-gastric variceal bleeding following endoscopic therapy for liver cirrhosis19.

The INR-ALB grading system successfully assessed rebleeding, particularly early rebleeding, in cirrhotic patients with EGVB following endoscopic therapy. 20.

These ALBI -associated scores have received a lot of attention and are considered potential alternatives to CTP and MELD as prognostic indicators in patients with liver cirrhosis. These objective scores are considered better predictors of liver decompensated events, especially in stratifying risk for portal hypertension 14,21 MELD 3.0 affords more accurate mortality prediction in general than MELD Na and addresses determinants of waitlist outcomes including the sex disparity 22.

A MELD 3.0 less than 12 was associated with less than 5 % mortality and >20 was associated with >20% mortality 23.

Secondary to drawbacks of CTP (evaluated subjectively) and MELD (complexity in its calculation) for prognosis of patients with variceal bleeding, ALBI -associated scores (ALBI, PALBI and INR-ALBI) could be rapid, effective, and validated scores in prediction the outcome of such patients and to identify candidates for an early transjugular intrahepatic porto-systemic shunt procedure.

ELIGIBILITY:
Inclusion Criteria:

* Any cirrhotic patients above the age of 18 years old of both sexes, present with variceal bleeding.

Exclusion Criteria:

* Patients with other causes of upper gastrointestinal bleeding (UGIB).
* Patients who are receiving anticoagulant or antiplatelet therapy.
* Patients with HCC, other malignant tumors, and hematological disease at the time of recruitment or during follow up.
* Patients who underwent transjugular intrahepatic portosystemic shunt, splenectomy, or partial splenic embolization.
* Patients with liver cirrhosis and portal vein thrombosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any cirrhotic patients present with variceal bleeding.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
assess the prognostic performance of the ALBI_associated scores and new MELD .3 in predicting the short-term outcomes of patients with cirrhosis presenting with acute variceal bleeding. | baseline
  assess the prognostic performance of the ALBI_associated scores (ALBI, PALBI and INR-ALBI score) and new MELD .3 in predicting the short-term outcomes (early re-bleeding and early mortality) of patients with cirrhosis presenting with acute variceal bleeding, comparable to the CTP and MELD and MELD Na scores.

REFERENCES:
- [Background] Alqahtani SA, Jang S. Pathophysiology and Management of Variceal Bleeding. Drugs. 2021 Apr;81(6):647-667. doi: 10.1007/s40265-021-01493-2. Epub 2021 Mar 12. PMID 33710585
- [Background] Drolz A, Ferlitsch A, Fuhrmann V. Management of Coagulopathy during Bleeding and Invasive Procedures in Patients with Liver Failure. Visc Med. 2018 Aug;34(4):254-258. doi: 10.1159/000491106. Epub 2018 Jul 16. PMID 30345282
- [Background] Reiberger T, Puspok A, Schoder M, Baumann-Durchschein F, Bucsics T, Datz C, Dolak W, Ferlitsch A, Finkenstedt A, Graziadei I, Hametner S, Karnel F, Krones E, Maieron A, Mandorfer M, Peck-Radosavljevic M, Rainer F, Schwabl P, Stadlbauer V, Stauber R, Tilg H, Trauner M, Zoller H, Schofl R, Fickert P. Austrian consensus guidelines on the management and treatment of portal hypertension (Billroth III). Wien Klin Wochenschr. 2017 Nov;129(Suppl 3):135-158. doi: 10.1007/s00508-017-1262-3. Epub 2017 Oct 23. PMID 29063233
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Sharara AI, Rockey DC. Gastroesophageal variceal hemorrhage. N Engl J Med. 2001 Aug 30;345(9):669-81. doi: 10.1056/NEJMra003007. No abstract available. PMID 11547722
- [Background] Johnson PJ, Berhane S, Kagebayashi C, Satomura S, Teng M, Reeves HL, O'Beirne J, Fox R, Skowronska A, Palmer D, Yeo W, Mo F, Lai P, Inarrairaegui M, Chan SL, Sangro B, Miksad R, Tada T, Kumada T, Toyoda H. Assessment of liver function in patients with hepatocellular carcinoma: a new evidence-based approach-the ALBI grade. J Clin Oncol. 2015 Feb 20;33(6):550-8. doi: 10.1200/JCO.2014.57.9151. Epub 2014 Dec 15. PMID 25512453
- [Background] Chan AW, Chan RC, Wong GL, Wong VW, Choi PC, Chan HL, To KF. New simple prognostic score for primary biliary cirrhosis: Albumin-bilirubin score. J Gastroenterol Hepatol. 2015 Sep;30(9):1391-6. doi: 10.1111/jgh.12938. PMID 25753927
- [Background] Elshaarawy O, Allam N, Abdelsameea E, Gomaa A, Waked I. Platelet-albumin-bilirubin score - a predictor of outcome of acute variceal bleeding in patients with cirrhosis. World J Hepatol. 2020 Mar 27;12(3):99-107. doi: 10.4254/wjh.v12.i3.99. PMID 32231763
- [Background] Li F, Wang T, Liang J, Qian B, Tang F, Gao Y, Lv J. Albumin-bilirubin grade and INR for the prediction of esophagogastric variceal rebleeding after endoscopic treatment in cirrhosis. Exp Ther Med. 2023 Sep 11;26(5):501. doi: 10.3892/etm.2023.12200. eCollection 2023 Nov. PMID 37822588
- [Background] Wang J, Zhang Z, Yan X, Li M, Xia J, Liu Y, Chen Y, Jia B, Zhu L, Zhu C, Huang R, Wu C. Albumin-Bilirubin (ALBI) as an accurate and simple prognostic score for chronic hepatitis B-related liver cirrhosis. Dig Liver Dis. 2019 Aug;51(8):1172-1178. doi: 10.1016/j.dld.2019.01.011. Epub 2019 Jan 26. PMID 30765220
- [Background] Kim WR, Mannalithara A, Heimbach JK, Kamath PS, Asrani SK, Biggins SW, Wood NL, Gentry SE, Kwong AJ. MELD 3.0: The Model for End-Stage Liver Disease Updated for the Modern Era. Gastroenterology. 2021 Dec;161(6):1887-1895.e4. doi: 10.1053/j.gastro.2021.08.050. Epub 2021 Sep 3. PMID 34481845
- [Background] Buckholz A, Wong R, Curry MP, Baffy G, Chak E, Rustagi T, Mohanty A, Fortune BE. MELD, MELD 3.0, versus Child score to predict mortality after acute variceal hemorrhage: A multicenter US cohort. Hepatol Commun. 2023 Sep 11;7(10):e0258. doi: 10.1097/HC9.0000000000000258. eCollection 2023 Oct 1. PMID 37695092
- [Background] Jairath V, Rehal S, Logan R, Kahan B, Hearnshaw S, Stanworth S, Travis S, Murphy M, Palmer K, Burroughs A. Acute variceal haemorrhage in the United Kingdom: patient characteristics, management and outcomes in a nationwide audit. Dig Liver Dis. 2014 May;46(5):419-26. doi: 10.1016/j.dld.2013.12.010. Epub 2014 Jan 14. PMID 24433997
- [Background] Boregowda U, Umapathy C, Halim N, Desai M, Nanjappa A, Arekapudi S, Theethira T, Wong H, Roytman M, Saligram S. Update on the management of gastrointestinal varices. World J Gastrointest Pharmacol Ther. 2019 Jan 21;10(1):1-21. doi: 10.4292/wjgpt.v10.i1.1. PMID 30697445
- [Background] Yang H, Pan C, Liu Q, Wang Y, Liu Z, Cao X, Lei J. Correlation between the Glasgow-Blatchford score, shock index, and Forrest classification in patients with peptic ulcer bleeding. Turk J Med Sci. 2020 Jun 23;50(4):706-712. doi: 10.3906/sag-1906-154. PMID 32041384
- [Background] van Dam GM, Gips CH, Reisman Y, Maas KW, Purmer IM, Huizenga JR, Verbaan BW. Major clinical events, signs and severity assessment scores related to actual survival in patients who died from primary biliary cirrhosis. A long-term historical cohort study. Hepatogastroenterology. 1999 Jan-Feb;46(25):108-15. PMID 10228773
- [Background] Shetty K, Rybicki L, Carey WD. The Child-Pugh classification as a prognostic indicator for survival in primary sclerosing cholangitis. Hepatology. 1997 May;25(5):1049-53. doi: 10.1002/hep.510250501. PMID 9141416
- [Background] Zhao Y, Ren M, Lu G, Lu X, Yin Y, Zhang D, Wang X, Ma W, Li Y, Cai G, Lin Y, He S. The Prognosis Analysis of Liver Cirrhosis with Acute Variceal Bleeding and Validation of Current Prognostic Models: A Large Scale Retrospective Cohort Study. Biomed Res Int. 2020 Aug 16;2020:7372868. doi: 10.1155/2020/7372868. eCollection 2020. PMID 32879889